CLINICAL TRIAL: NCT05406284
Title: A Novel Coronary Bifurcation Stenting Technique With Minimal Protrusion: Double Kissing Nano-Culotte Stenting
Brief Title: DK Nano-Culotte Stenting For Coronary Bifurcation Lesion
Status: Recruiting | Type: Observational
Sponsor: Istanbul Mehmet Akif Ersoy Educational and Training Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: IMAEETH-3
Record Dates: First submitted 2022-06-01; First posted 2022-06-06 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Coronary Artery Disease
Keywords: coronary bifurcation lesion; DK nano-culotte stenting
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- double kissing nano culotte stenting
  Interventions: Procedure: double kissing nano culotte stenting

INTERVENTIONS:
Procedure: double kissing nano culotte stenting — patients with true coronary bifurcation lesion treating with double kissing nano culotte stunting technique

SUMMARY:
True coronary bifurcation lesions are still great of interest due to their complex anatomy, uncertainty of optimal stenting strategy and increased adverse cardiovascular outcomes. Provisional stenting is recommended in patients with non-complex coronary lesions while 2-stent strategies should be considered in complex coronary bifurcation lesions. However, optimal 2-stent strategy is still controversial. Double kissing (DK) crush stenting is the prominent technique in true bifurcation lesion, especially in patients with left main coronary artery disease. DK mini-culotte stenting, increasing use in clinical practice, has become popular over DK crush stenting. It was demonstrated in a bench test that stent malapposition was lower in the DK mini-culotte stenting compared to the DK crush technique. Thus, DK mini-culotte stenting may be preferred over DK crush stenting in complex true coronary bifurcation lesion. On the other hand, it was demonstrated in previous studies, less than minimal protrusion (generally called as nano protrusion) had better clinical outcomes. Kawasaki et al was first demonstrated the minimal (nano) protrusion of culotte stenting technique. Then, Toth et al revealed a novel modified culotte stenting technique named single string culotte. There was no major adverse cardiac events (MACE) in patients underwent single string stenting technique with a median follow-up period of 6±4 months. Unsurprisingly there was no MACE occurred in patients who underwent Szabo 2-stent technique. In the light of foregoing data, the least possible amount of protrusion is known to have the best results. In addition to this, double kissing balloon dilatation with culotte stenting technique seems to have better results than other stenting techniques. In our study, we aimed to evaluate the angiographic and clinical results of a novel DK Nano-Culotte stenting in coronary bifurcation lesion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with de novo true bifurcation lesion (Medina classification 1,1,1 or 0,1,1 or 1,0,1)
* The main vessel diameter is least 2.5 mm and the side branch diameter is at least 2.25 mm

Exclusion Criteria:

* Patients presenting with ST segment elevation myocardial infarction, cardiogenic shock and Killip class III-IV heart failure
* Patients with a history of coronary artery bypass grafting surgery
* Patients with a chronic total occlusion in the bifurcation area
* Lesions with severe calcification that needs additional intervention such as atherectomy
* Patients who are not suitable to use long term dual antiplatelet therapy and patients not participating in clinical follow-up
* Patients with hematological disorders, malignancy, end stage renal (GFR<30 ml/min) and hepatic failure
* Patients with active bleeding
* Pregnant women
* Patients with life-expectancy < 1 year
* Patients treated with small open cell stent platforms

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with stable or unstable angina pectoris or patients with non-ST segment elevation myocardial infarction undergoing percutaneous coronary intervention and performing DK nano culotte stunting technique
Sampling Method: Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
MACE (major adverse cardiovascular events) | 6 months
  target vessel revascularization, myocardial infarction or cardiac death

SECONDARY OUTCOMES:
MACCE (major adverse cerebral and cardiovascular events) | 6, 12 months
  all cause death, myocardial infarction, target vessel revascularization, in-stent thrombosis/restenosis or stroke
target lesion failure | 6, 12 months
  target lesion revascularization, myocardial infarction, cardiac death

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Mehmet Akif Ersoy Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Steigen TK, Maeng M, Wiseth R, Erglis A, Kumsars I, Narbute I, Gunnes P, Mannsverk J, Meyerdierks O, Rotevatn S, Niemela M, Kervinen K, Jensen JS, Galloe A, Nikus K, Vikman S, Ravkilde J, James S, Aaroe J, Ylitalo A, Helqvist S, Sjogren I, Thayssen P, Virtanen K, Puhakka M, Airaksinen J, Lassen JF, Thuesen L; Nordic PCI Study Group. Randomized study on simple versus complex stenting of coronary artery bifurcation lesions: the Nordic bifurcation study. Circulation. 2006 Oct 31;114(18):1955-61. doi: 10.1161/CIRCULATIONAHA.106.664920. Epub 2006 Oct 23. PMID 17060387
- [Background] Colombo A, Bramucci E, Sacca S, Violini R, Lettieri C, Zanini R, Sheiban I, Paloscia L, Grube E, Schofer J, Bolognese L, Orlandi M, Niccoli G, Latib A, Airoldi F. Randomized study of the crush technique versus provisional side-branch stenting in true coronary bifurcations: the CACTUS (Coronary Bifurcations: Application of the Crushing Technique Using Sirolimus-Eluting Stents) Study. Circulation. 2009 Jan 6;119(1):71-8. doi: 10.1161/CIRCULATIONAHA.108.808402. Epub 2008 Dec 22. PMID 19103990
- [Background] Hildick-Smith D, de Belder AJ, Cooter N, Curzen NP, Clayton TC, Oldroyd KG, Bennett L, Holmberg S, Cotton JM, Glennon PE, Thomas MR, Maccarthy PA, Baumbach A, Mulvihill NT, Henderson RA, Redwood SR, Starkey IR, Stables RH. Randomized trial of simple versus complex drug-eluting stenting for bifurcation lesions: the British Bifurcation Coronary Study: old, new, and evolving strategies. Circulation. 2010 Mar 16;121(10):1235-43. doi: 10.1161/CIRCULATIONAHA.109.888297. Epub 2010 Mar 1. PMID 20194880
- [Background] Ferenc M, Gick M, Kienzle RP, Bestehorn HP, Werner KD, Comberg T, Kuebler P, Buttner HJ, Neumann FJ. Randomized trial on routine vs. provisional T-stenting in the treatment of de novo coronary bifurcation lesions. Eur Heart J. 2008 Dec;29(23):2859-67. doi: 10.1093/eurheartj/ehn455. Epub 2008 Oct 9. PMID 18845665
- [Background] Chen SL, Zhang JJ, Han Y, Kan J, Chen L, Qiu C, Jiang T, Tao L, Zeng H, Li L, Xia Y, Gao C, Santoso T, Paiboon C, Wang Y, Kwan TW, Ye F, Tian N, Liu Z, Lin S, Lu C, Wen S, Hong L, Zhang Q, Sheiban I, Xu Y, Wang L, Rab TS, Li Z, Cheng G, Cui L, Leon MB, Stone GW. Double Kissing Crush Versus Provisional Stenting for Left Main Distal Bifurcation Lesions: DKCRUSH-V Randomized Trial. J Am Coll Cardiol. 2017 Nov 28;70(21):2605-2617. doi: 10.1016/j.jacc.2017.09.1066. Epub 2017 Oct 30. PMID 29096915
- [Background] Toth GG, Sasi V, Franco D, Prassl AJ, Di Serafino L, Ng JCK, Szanto G, Schneller L, Ang HY, Plank G, Wijns W, Barbato E. Double-kissing culotte technique for coronary bifurcation stenting. EuroIntervention. 2020 Oct 9;16(9):e724-e733. doi: 10.4244/EIJ-D-20-00130. PMID 32338608
- [Background] Kawasaki T, Koga H, Serikawa T. Modified culotte stenting technique for bifurcation lesions: the cross-stenting technique. J Invasive Cardiol. 2010 May;22(5):243-6. PMID 20440044
- [Background] G Toth G, Pyxaras S, Mortier P, De Vroey F, Di Gioia G, Adjedj J, Pellicano M, Ferrara A, De Schryver T, Van Hoorebeke L, Verhegghe B, Barbato E, De Bruyne B, De Beule M, Wijns W. Single String Technique for Coronary Bifurcation Stenting: Detailed Technical Evaluation and Feasibility Analysis. JACC Cardiovasc Interv. 2015 Jun;8(7):949-59. doi: 10.1016/j.jcin.2015.01.037. Epub 2015 May 20. PMID 26003016
- [Background] Yang H, Qian J, Huang Z, Ge J. Szabo 2-stent technique for coronary bifurcation lesions: procedural and short-term outcomes. BMC Cardiovasc Disord. 2020 Jul 7;20(1):325. doi: 10.1186/s12872-020-01605-y. PMID 32635890